CLINICAL TRIAL: NCT05322889
Title: Prevention of Paclitaxel-induced Neuropathic Pain by Telmisartan in Patients With Planned Paclitaxel Chemotherapy Due to Ovarian or Breast Cancer (PrevTel)
Brief Title: Prevention of Paclitaxel-induced Neuropathic Pain in Patients With Planned Paclitaxel Chemotherapy (PrevTel)
Acronym: PrevTel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Frank Behrens (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Frank Behrens, Head of clinical research - Representative of the Sponsor, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TMP-0315-2018
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Neuropathic Pain; Chemotherapy Effect
Keywords: chemotherapy induced peripheral neuropathic pain, breast cancer; ovarian cancer; paclitaxel
MeSH Terms: conditions — Neuralgia; Breast Neoplasms; Ovarian Neoplasms | interventions — Telmisartan

STUDY DESIGN:
Intervention Model Description: monocentric, open label, single-arm trial
Masking Description: no blinding necessary
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with Telmisartan (Experimental): Telmisartan (open), 80 mg daily p.o. (after run-in phase with 40 mg for 7 days).
  for 12 weeks
  Interventions: Drug: Telmisartan tablets

INTERVENTIONS:
Drug: Telmisartan tablets — 12 weeks treatment

SUMMARY:
Phase IIa clinical trial will be conducted with patients requiring in-label paclitaxel-chemotherapy due to ovarian or breast cancer. The efficacy of a 12-week telmisartan treatment, starting one week before planned paclitaxel-administration to prevent PIPNP (paclitaxel-induced peripheral neuropathic pain) will be assessed by measurement of occurrence of clinical symptoms of PIPNP as well as lipid profiles

DETAILED DESCRIPTION:
Paclitaxel is a cytostatic drug that is widely used for the first-line treatment of breast- and ovarian cancer and causes neuropathic pain in up to 87% of treated patients Treating mice with telmisartan causes a strong reduction of PIPNP, thus indicating that telmisartan may be a promising pharmacological treatment option for PIPNP in patients. It is proposed that telmisartan reduces the inflammatory component of PIPNP.

Telmisartan has a good risk profile, low occurrence of side effects and is generally well tolerated in patients.These collective characteristics make it a suitable, already approved and appropriate substance for combination therapy with paclitaxel.

Therefore, telmisartan is a promising candidate to potentially prevent PIPNP in patients whose safety profile is well known due to preclinical and clinical trials for the indication of hypertension and coronary heart disease. Moreover, due to its mechanisms it might as well reduce symptoms of PIPNP sufficiently without severe side effects.

To validate these observations clinically, this phase IIa clinical trial will be conducted with breast and ovarian cancer patients requiring in-label paclitaxel-chemotherapy. The efficacy of a 12-week telmisartan treatment initiated before the first administration of paclitaxel to prevent PIPNP will be assessed.

Moreover, beside lipid profiles, quantitative sensoric testing of pain characteristics in focus on biomarker detection and development that may be useful for a precision medicine approach will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ovarian or breast cancer who are clinically eligible for paclitaxel therapy and for whom paclitaxel chemotherapy is planned (with use of standard treatment) in clinical routine care.
* Female patients ≥ 18 years and ≤ 80 years
* The patient must have completed radiotherapy or surgery for central nervous system (CNS) metastases > 2 weeks prior to screening (SCR). Patients must be neurologically stable, having no new neurological deficits on clinical examination, and no new findings on CNS imaging as documented in clinical routine care. If patients require steroids for management of CNS metastases, they must have been on a stable dose of steroids for 2 weeks preceding SCR.
* Written informed consent obtained prior to the initiation of any protocol-required procedures
* Willingness to comply to study procedures and study protocol

Exclusion Criteria:

* Previously diagnosed or current peripheral neuropathic pain
* Other severe pain that might impair the assessment of neuropathic pain
* DN4 score ≥ 4
* Previous chemotherapy (incl. paclitaxel) within the last 5 years (treatment with cyclophosphamide and an anthracycline as part of an ongoing adjuvant or neo-adjuvant regimen is allowed)
* Current or planned combinational chemotherapy-regimens, e.g., with platinum-based drugs (Her2 antibodies are allowed; paclitaxel combination with trastuzumab +/- pertuzumab is allowed)
* All primary central nervous system (CNS) tumors or symptomatic CNS metastases that are neurologically unstable (Note: Only patients with controlled CNS metastases may participate in this trial)
* Previously reported intolerance to Angiotensin II (AT1) -receptor-blockers
* Hypotension (blood pressure < 110/70 mmHg; median from 3 measurements; start of measurement after patients has been seated for at least 5 minutes)
* Current intake of aliskiren, digoxin or Angiotensin-converting-enzyme (ACE)-inhibitors at baseline (BL) (treatment change from ACE-inhibitors to telmisartan is allowed, with treatment start of telmisartan at BL)
* Current intake of antidepressants (e.g., amitriptylin), antiepileptics (e.g., gabapentin, pregabalin, lamotrigine), duloxetine, glutamin, vitamin E
* Current intake of telmisartan at SCR
* Insufficient hepatic or renal function at SCR:

  * Serum creatinine ≥ 1.5 x upper limit of normal (ULN)
  * Total bilirubin > 1.5 x ULN
  * Glutamate-Oxalacetete-Transaminase/Glutamate-Pyruvate-Transaminase (GOT/GPT) ≥ 3 x ULN or >5 in case of documented liver metastasis
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* History of or current severe psychological illness or condition
* Uncontrolled coronary angina or symptomatic congestive heart failure (NYHA (New York Heart Association) Class III or IV)
* Patients with current malignant disease, other than that being treated in this study. Exceptions to this exclusion criterion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to SCR; completely resected basal cell and squamous cell skin cancers; and completely resected carcinoma in situ of any type
* Evidence of significant uncontrolled concomitant diseases or serious and/or uncontrolled diseases that are likely to interfere with the evaluation of the patient's safety and of the study outcome
* History of or evidence of current active Hepatitis B or C or Human Immunodeficiency Virus (HIV) infection with documentation not older than 8 weeks (due to blood sample processing for lipid profile analysis)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
efficacy of telmisartan to prevent new onset of Paclitaxel- induced peripheral neuropathic pain (PIPNP) | week 12
  Proportion of patients without onset of PIPNP measured by median Quality of life questionaire (doleur neuropathic questionnaire) DN4, DN4 < 4

SECONDARY OUTCOMES:
Proportion of patients with new onset of PIPNP | Day 14
  Douleur Neuropathique 4 (DN4) questionnaire (DN4 ≥ 4) higher score means more pain, minimum 0 to maximum 10 points
Proportion of patients with new onset of PIPNP | Day 28
  DN4 questionnaire (DN4 ≥ 4) higher score means more pain, minimum 0 to maximum 10 points
Proportion of patients with new onset of PIPNP | Day 49
  DN4 questionnaire (DN4 ≥ 4) higher score means more pain, minimum 0 to maximum 10 points
Proportion of patients with new onset of PIPNP | Day 70
  DN4 questionnaire DN4 ≥ 4
Proportion of patients with new onset of PIPNP | Day 84
  DN4 questionnaire DN4 ≥ 4 higher score means more pain, minimum 0 to maximum 10 points
Change of pain intensity to baseline - Paindetect | Day 14
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain intensity to baseline - Paindetect | Day 28
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain intensity to baseline - Paindetect | Day 49
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain intensity to baseline - Paindetect | Day 70
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain intensity to baseline - Paindetect | Day 84
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain intensity to baseline - VAS | Day 14
  patient global pain visual analogue scale (VAS-Pain), minimum 0 to 10, higher score means more pain
Change of pain intensity to baseline - VAS | Day 28
  patient global pain visual analogue scale (VAS-Pain), minimum 0 to 10, higher score means more pain
Change of pain intensity to baseline - VAS | Day 49
  patient global pain visual analogue scale (VAS-Pain), minimum 0 to 10, higher score means more pain
Change of pain intensity to baseline - VAS | Day 70
  patient global pain visual analogue scale (VAS-Pain), minimum 0 to 10, higher score means more pain
Change of pain intensity to baseline - VAS | Day 84
  patient global pain visual analogue scale (VAS-Pain), minimum 0 to 10, higher score means more pain
Change in pain pattern to baseline | Day 14
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change in pain pattern to baseline | Day 28
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change in pain pattern to baseline | Day 49
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change in pain pattern to baseline | Day 70
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change in pain pattern to baseline | Day 84
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain quality to baseline | Day 14
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain quality to baseline | Day 28
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain quality to baseline | Day 49
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain quality to baseline | Day 70
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change of pain quality to baseline | Day 84
  PainDetect questionnaire, higher score means more pain, minimum 0 to 38 maximum
Change in quality of life (QoL) to baseline | Day 14
  Functional Assessment of Cancer Therapy/Gynecologic Oncology (FACT/ GOG-NTX), 38 items questionaire each to be scored from 0 (Not at all) to 4 (Very much) - total score could be between 0 and 152 Group-Neurotoxicity (FACT/GOG-NTX questionnaire) - some items are reverse scored. Subscale scores, total scores possible
Change in quality of life (QoL) to baseline | Day 49
  Functional Assessment of Cancer Therapy/Gynecologic Oncology (FACT/ GOG-NTX), 38 items questionaire each to be scored from 0 (Not at all) to 4 (Very much) - total score could be between 0 and 152 Group-Neurotoxicity (FACT/GOG-NTX questionnaire) - some items are reverse scored. Subscale scores, total scores possible
Change in quality of life (QoL) to baseline | Day 28
  Functional Assessment of Cancer Therapy/Gynecologic Oncology (FACT/ GOG-NTX), 38 items questionaire each to be scored from 0 (Not at all) to 4 (Very much) - total score could be between 0 and 152
Change in quality of life (QoL) to baseline | Day 70
  Functional Assessment of Cancer Therapy/Gynecologic Oncology (FACT/ GOG-NTX), 38 items questionaire each to be scored from 0 (Not at all) to 4 (Very much) - total score could be between 0 and 152
Change in quality of life (QoL) to baseline | Day 84
  Functional Assessment of Cancer Therapy/Gynecologic Oncology (FACT/ GOG-NTX), 38 items questionaire each to be scored from 0 (Not at all) to 4 (Very much) - total score could be between 0 and 152
cumulative incidence of neuropathic pain | throughout study treatment - 12 weeks
  documented by physician
Quantification of the incidence of paclitaxel-associated acute pain syndrome (PAPS) | throughout study treatment - 12 weeks
  documented by physician
proportion of patients in need of PIPNP symptomatic therapy | throughout study treatment - 12 weeks
  determined by treating physician - documented in case report form
Assessment of frequency of adverse events | throughout study treatment - 12 weeks
  determined by using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Assessment of severity of adverse events | throughout study treatment - 12 weeks
  determined by using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Assessment relatedness of adverse events | throughout study treatment - 12 weeks
  determined by using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Assessment of type of adverse events | throughout study treatment - 12 weeks
  determined by using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sebastian, MD, Principal Investigator — Department of Haematology/Medical Onkology, University Hospital, Goethe-University Frankfurt
Locations (1):
- Department of Haematology/Medical Onkology, University Hospital, Goethe-University Frankfurt, Frankfurt, Germany